CLINICAL TRIAL: NCT03349424
Title: A Multi-center, Randomized, Controlled Study: Somatostatin Prevent Post-operation Pancreatic Fistula (POPF) in Intermediate Risk Patients After Pancreaticoduodenectomy
Brief Title: Somatostatin Prevent Post-operation Pancreatic Fistula in Intermediate Risk Patients After Pancreaticoduodenectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, zhang taiping, Deputy Director,Professor,Chief Physician of General Surgery Department, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS200115_0006
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Fistula
Keywords: Somatostatin; Pancreatic Fistula; Intermediate Risk; Pancreaticoduodenectomy
MeSH Terms: conditions — Pancreatic Fistula | interventions — Somatostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stilamin group (Experimental): Patients in the Stilamin group will be continuous intravenous infusion with the somatostatin in addition to postoperative conventional treatment.
  Interventions: Drug: Somatostatin
- Control group (No Intervention): Patients in the control group will receive the postoperative conventional treatment, without addition of any new medicines.

INTERVENTIONS:
Drug: Somatostatin — Patients in the Stilamin group will be continuous intravenous infusion with the somatostatin (Stilamin®) of 250μg/h, beginning within 3 hours (Visit 1) after the operation and lasting for 120 hours (each subject will receive the Stilamin of 30mg in total), and other postoperative conventional treatment protocol remain unchanged.
  Other Names: Stilamin
  Arms: Stilamin group

SUMMARY:
This study is designed to assess the preventive effects of somatostatin on post-operation pancreatic fistula in intermediate risk patients after pancreaticoduodenectomy. Patients assigned into the treatment group will be continuous intravenous infusion with the somatostatin (Stilamin®) in addition to conventional treatments (including infection prevention, nutrition support and acid suppression therapy, etc.).The pancreatic fistula incidence will be monitored within 30 days after operation.

DETAILED DESCRIPTION:
This is a multi-center randomized, controlled clinical trial. A total of 200 patients are expected to be recruited. Each trial center recruits subjects based on the sequential principle and inspect the inclusion and exclusion criteria after PD and subjects meeting the standard are assigned randomly to the treatment group or control group. Apart from conventional treatments (including infection prevention, nutrition support and acid suppression therapy, etc.), the treatment group will be continuous intravenous infusion with the somatostatin (Stilamin®) of 250μg/h for 120h (total dose of 6mg/day x 5 days=30mg), beginning within 3 hours after the operation; the control group will accept conventional treatments other than the Stilamin.

The pancreatic fistula incidence, biochemical leak incidence, morbidity and number of other complications related to the pancreatectomy, length of stay in hospital, hospitalization cost, re-admission rate and re-operation rate will be monitored within 30 days after operation. Subjects will be visited for 5 times from the start to the end of the study.

Statistical Methods:Number of patients who had pancreatic fistula after surgery will be analyzed using Chi-square test.Secondary endpoints: Continuous variates will be described as mean± SD; attempted to be analyzed using analysis of variance. Categorical variates will be described as rate; attempted to be analyzed using Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 year
2. Patients underwent pancreaticoduodenectomy
3. Fistula Risk Score recommended by ISGPS is intermediate risk
4. Inform consent obtained

Exclusion Criteria:

1. Pervious pancreatic surgery history
2. Received somatostatin or analogues treatment less than 5 half-life periods before surgery
3. Known allergy to somatostatin or mannitol
4. Woman who is pregnant, plan to be pregnant or during lactation period
5. Attended other clinical trials within 30 days
6. All contraindications to somatostatin (Stilamin®)
7. Patients with any serious disease that investigator considers he/she should be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Incidence of post-operative pancreatic fistula | 30 days after operation
  A clinically relevant postoperative pancreatic fistula is now defined as a drain output of any measurable volume of fluid with an amylase level >3 times the upper limit of institutional normal serum amylase activity, associated with a clinically relevant development/condition related directly to the postoperative pancreatic fistula.

CONTACTS AND LOCATIONS:
Overall Officials: Yupei Zhao, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Study Group of Pancreatic Surgery in Chinese Society of Surgery of Chinese Medical Association; Pancreatic Disease Committee of Chinese Research Hospital Association; Editorial Board of Chinese Journal of Surgery. [A consensus statement on the diagnosis, treatment, and prevention of common complications after pancreatic surgery (2017)]. Zhonghua Wai Ke Za Zhi. 2017 May 1;55(5):328-334. doi: 10.3760/cma.j.issn.0529-5815.2017.05.003. Chinese. PMID 28464570
- [Background] Callery MP, Pratt WB, Kent TS, Chaikof EL, Vollmer CM Jr. A prospectively validated clinical risk score accurately predicts pancreatic fistula after pancreatoduodenectomy. J Am Coll Surg. 2013 Jan;216(1):1-14. doi: 10.1016/j.jamcollsurg.2012.09.002. Epub 2012 Nov 2. PMID 23122535
- [Background] Gouillat C, Chipponi J, Baulieux J, Partensky C, Saric J, Gayet B. Randomized controlled multicentre trial of somatostatin infusion after pancreaticoduodenectomy. Br J Surg. 2001 Nov;88(11):1456-62. doi: 10.1046/j.0007-1323.2001.01906.x. PMID 11683740
- [Derived] Cao Z, Qiu J, Guo J, Xiong G, Jiang K, Zheng S, Kuang T, Wang Y, Zhang T, Sun B, Qin R, Chen R, Miao Y, Lou W, Zhao Y. A randomised, multicentre trial of somatostatin to prevent clinically relevant postoperative pancreatic fistula in intermediate-risk patients after pancreaticoduodenectomy. J Gastroenterol. 2021 Oct;56(10):938-948. doi: 10.1007/s00535-021-01818-8. Epub 2021 Aug 28. PMID 34453212